CLINICAL TRIAL: NCT02128789
Title: Bring Communities and Technology Together for Healthy Aging
Acronym: ElderTree
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2013-0171; 5P50HS019917-04 (AHRQ); HS019917 (Other: Study Team)
Record Dates: First submitted 2014-03-26; First posted 2014-05-01 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: 65 Years Older; Requires IADL Support; Past Year History of Falls and/or Hospitalization
Keywords: Older Adults; Caregivers; Aging; Support

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Condition (No Intervention): Subjects receive usual care and support. No study intervention provided
- Elder Tree Condition (Experimental): Elder Tree website. Subjects receive usual care, support and access to the study intervention website.
  Interventions: Other: Elder Tree website

INTERVENTIONS:
Other: Elder Tree website — Elder Tree is a private, secure information, support and communication website developed for this study.
  Arms: Elder Tree Condition

SUMMARY:
Technology has been created to help older adults age well in their homes, but adoption and acceptance have been slow. The researchers are developing a low-cost web-based technology, called Elder Tree, for older adults and caregivers to address key challenges older adults face, such as loneliness and isolation, falls, loss of driving privileges, relapsing from proven falls prevention strategies, and unreliable home services. Elder Tree is being developed and tested with older adults and caregivers to identify, 1) usability issues such as font size, navigation and interface (audio, video,text) and 2) content and tailoring issues such as identifying local resources and events. This study will employ a randomized longitudinal design comparing a control group to an intervention group over a 12-month period. Investigators hypothesize that older adults using Elder Tree will experience greater independence and quality of life when compared to the control group. Investigators will use quantitative measures to determine how much our intervention improves: quality of life and health system use. These measures will help us to determine the cost effectiveness of Elder Tree. Investigators will recruit and test Elder Tree in 3 Regional Aging and Disability Resource Centers; one urban, one suburban and one rural setting, so to account for environmental and community differences. The older adult and their caregiver will be randomized to the same treatment group. Investigators will measure the effect over the 12 month intervention period and a 6 month follow-up period at 18 months.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* In need of IADL support
* 1 years history or risk of hospitalization or falls
* Resident of the following counties Milwaukee, WI, Waukesha Wi or Richland County
* Must be able to read English at a 6th grade level.

Exclusion Criteria:

* Under 65 years of age
* Unable to read English
* Not a resident of the above listed counties.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of older adult subjects with increased independence and quality of life from baseline to 18 months | Change in independence and quality of life will be assessed at 6, 12 , 18 months
  Compared to the control group elders using Elder Tree will experience greater independence and quality of life and will have fewer unscheduled clinical and emergency room visits and hospital and nursing home stays.

SECONDARY OUTCOMES:
Number of caregiver subjects with improved satisfaction | Change in improved caregiver satisfaction will be assessed at 6, 12 , 18 months
  Compared to the control group, caregivers using Elder Tree will experience improved satisfaction, coping and appraisal.

CONTACTS AND LOCATIONS:
Locations (1):
- University of WI Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Gustafson DH Sr, Kornfield R, Mares ML, Johnston DC, Cody OJ, Yang EF, Gustafson DH Jr, Hwang J, Mahoney JE, Curtin JJ, Tahk A, Shah DV. Effect of an eHealth intervention on older adults' quality of life and health-related outcomes: a randomized clinical trial. J Gen Intern Med. 2022 Feb;37(3):521-530. doi: 10.1007/s11606-021-06888-1. Epub 2021 Jun 7. PMID 34100234
- [Derived] Gustafson DH Sr, McTavish F, Gustafson DH Jr, Mahoney JE, Johnson RA, Lee JD, Quanbeck A, Atwood AK, Isham A, Veeramani R, Clemson L, Shah D. The effect of an information and communication technology (ICT) on older adults' quality of life: study protocol for a randomized control trial. Trials. 2015 Apr 25;16:191. doi: 10.1186/s13063-015-0713-2. PMID 25909465